CLINICAL TRIAL: NCT03046888
Title: ROBOTIC PYELOLITHIOTOMY VERSUS PERCUTANEOUS NEPHROLITHOTOMY (PCNL).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Chief Urologist, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-598
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Prospectively randomized study in patients with renal pelvic stones who are candidate to standard PCNL procedure. One to one, controlled clinical trial. Patients will be randomly allocated into two groups, 20 patients in each group. Group A will be scheduled to receive routine standard PCNL. Group B will be scheduled to receive RP.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCNL (Experimental): Percutant nephrolithotomy is a standard procedure for stones treatment over 2 cm.The puncture will be performed with an 18-G nephrostomy needle. The access thus gained guaranteed the transpapillary route of the percutaneous tract, a basic condition for the prevention of bleeding. Subsequently, following withdrawal of the puncture needle and urine drainage, a flexible guidewire will be inserted and advanced to the upper calyx or ureter.
  Interventions: Procedure: Robot assisted pyelolithotomy
- Robot assisted pyelolithotomy (Experimental): Robot assisted pyelolithotomy, is a new technique to remove stones of more than 2 cm. A 12-mm camera port is placed at the level of the umbilicus and lateral. Two 8-mm robotic trocars are placed under direct vision and a 12-mm assistant port is placed in the midline a 5-8 cm above the umbilicus. After reflecting the colon medially, the renal pelvis will be dissected and identified, a flexible cystoscope will be inserted via an assisted trocar and introduced into the renal pelvis through a minor incision. The kidney stones will then be extracted with a basket and either removed via the port or placed in a specimen retrieval bag.
  Interventions: Procedure: Robot assisted pyelolithotomy

INTERVENTIONS:
Procedure: Robot assisted pyelolithotomy — A 12-mm camera port is placed at the level of the umbilicus and lateral; this port is moved farther laterally in morbidly obese patients to allow for the instruments to reach the target organs. Two 8-mm robotic trocars are placed under direct vision and a 12-mm assistant port is placed in the midline a 5-8 cm above the umbilicus. For right-sided stones, an additional 5-mm port is placed in the midline just below the xiphoid process for liver retraction. Placement of the trocars can be changed according to surgeon preference. After reflecting the colon medially, the renal pelvis will be dissected and identified, a flexible cystoscope will be inserted via an assisted trocar and introduced into the renal pelvis through a minor incision. The kidney stones will then be extracted with a basket and either removed via the port or placed in a specimen retrieval bag.

SUMMARY:
Prospectively randomized study in patients with renal pelvic stones who are candidate to standard PCNL procedure. One to one, controlled clinical trial. Patients will be randomly allocated into two groups, 20 patients in each group. Group A will be scheduled to receive routine standard PCNL. Group B will be scheduled to receive Robot assisted pyelolethotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Renal stones ≥2 cm.
3. Patients are candidate to PCNL.
4. Patient with ECOG performance score of 2 and less.
5. Able to give informed consent
6. Able to discharges home at the same day.

Exclusion Criteria:

1. Renal stones < 2cm and can managed by another technique.
2. Known with psychological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Postoperative hospital stay | 30 days
  the length of hospital stay efter each procedure

SECONDARY OUTCOMES:
Stones free rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No